CLINICAL TRIAL: NCT00239135
Title: An Open-label, Dose Escalation, Cohort Study to Determine the Maximum Tolerated Dose and Safety of PEP005 Topical Gel When Applied on Day 1 and Day 2 to Actinic Keratoses on the Shoulders, Chest, Back or Arms Followed by a Post-Treatment Follow-up Period Lasting at Four Weeks
Brief Title: Study to Determine the Maximum Tolerated Dose and Safety of PEP005 Topical Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-004
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Keratosis
Keywords: Actinic Keratosis; Topical; Maximum Tolerated Dose; Solar Keratosis; Sun Spots; Dermatology
MeSH Terms: conditions — Keratosis; Keratosis, Actinic; Melanosis | interventions — 3-ingenyl angelate

INTERVENTIONS:
Drug: PEP005

SUMMARY:
The purpose of this study is :

* To determine the maximum tolerated dose (MTD) for PEP005 Topical Gel in patients with actinic keratoses.
* To evaluate patients for clinical safety
* To determine the systemic absorption of PEP005 Topical Gel

DETAILED DESCRIPTION:
Actinic keratoses (AK) is a common skin condition characterized by rough, scaly patches or sores on the top layer of the skin which if left untreated can progress to skin cancer. Current treatments can cause scarring and hypopigmentation, be inconvenient, or require long treatment duration. Non-invasive alternative therapy for treatment of AK lesions is thus being researched.

This is an open label, dose escalation, cohort study to determine the maximum tolerated dose (MTD) of PEP005 Topical Gel, administered once daily for two consecutive days (90 ul gel applied topically over a 3 x 3cm template surrounding a target lesion), to patients with actinic keratoses (AK). The study will be conducted in one centre in the US. Three patients will be entered initially at the lowest dose level (0.01%) with up to an additional three patients to be entered in the event of a dose limiting toxicity (DLT) in the initial patients. DLT are defined as 'severe' local skin reactions observed by the Investigator, either prior to treatment on Day 2 ( following treatment on Day 1 ) or observed on Day 8 (following treatment on Day 2). Based on findings from phase I studies and the low systemic absorption found in non-clinical toxicokinetic evaluations, no systemic toxicity is anticipated.Once determined A total of 10 patients will be treated at the MTD in order to confirm it's determination. Based on findings from the phase I study, the starting dose will be 0.01% PEP005 Gel.

Secondary objectives of the study are (1) evaluate the clinical efficiency of PEP005 Topical Gel, when administered once daily for two consecutive days and (2) determine the systemic absorption of PEP005 Topical Gel at the MTD . Hematologic and biochemical assessments will be undertaken at the screening visit and at days 8 and 29 . Adverse events will be assessed at every study visit. Clinical response to treatment will be assessed at Days 8, 15 and 29.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* One AK lesion selected for treatment on the shoulders, chest, back or arms
* Longest diameter of the selected lesion between 3mm and 15mm
* Screening laboratory values within the references ranges as defined by the laboratory or "out of range" test results that are clinically acceptable to the Investigator
* Ability to follow study instructions and likely to complete all study requirements
* Written informed consent has been obtained
* Written Authorization for the Use and Release of Health and Research Study Information has been obtained
* Agreement from the patient to allow photographs of the selected lesion to be taken and used as part of the study data package.

Exclusion Criteria:

* Females of child bearing potential (a female is considered to be of childbearing potential unless she is post-menopausal, i.e no menses for at least 12 consecutive months or is without a uterus)
* Actinic Keratoses selected for treatment that are hypertrophic
* Location of the selected actinic keratoses lesion:

  1. within 5 cm of a scar
  2. within 5 cm of any actinic keratosis lesion not selected for treatment
  3. within 5 cm of an incompletely healed wound
  4. on the breast
  5. within 5 cm of an area previously treated with surgical excision
* Presence of suspected basal cell carcinoma or squamous cell carcinoma within 5 cm of the selected treatment area
* Presence of known or suspected metastatic disease
* History or evidence of skin conditions other than AK which would interfere with the evaluation of the study medication (e.g eczema, unstable psoriasis, xeroderma pigmentosa)
* Known sensitivity to any of the ingredients in the study medication
* A cosmetic or therapeutic procedure (e.g liquid nitrogen, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) located within 10cm of the actinic keratosis lesion selected for treatment during three months prior to study entry or anticipated treatment within 10cm of the selected lesion during the study
* Within four weeks prior to study entry, a cosmetic or therapeutic procedure located anywhere on the body
* Within three months prior to the study entry, treatment with 5-flourouracil, imiquimod, diclofenac, masoprocol, or photodynamic therapy for lesions located within 10cm of the actinic keratosis lesion selected for treatment
* Within four weeks prior to study entry, treatment with 5-flourouracil, imiquimod, masoprocol, or photodynamic therapy for lesion located anywhere on the body
* Previous treatment with other immunomodulators (e.g vinblastine, podophyllin, colhamin, camptothecin), cytotoxic drugs (e;g cyclophosphamide, azathioprine, chlorambucil, nitrogen mustard, methotrexate), or interferon/interferon inducers (other than imiquimod)within four weeks prior to study entry
* Previous treatment with psoralen plus UVA or use of UVB therapy within six months prior to study entry
* Patients who require or desire excess or prolonged exposure to ultraviolet light(e.g sunlight, tanning beds) during the study
* Use of medications that suppress the immune system within four weeks prior study entry (e.g cyclosporine, prednisone, methotrexate, alefacept, infliximab)
* Within four weeks prior to study entry, use of topical retinoids or light chemical peels located within 10cm of the actinic keratosis lesion selected for treatment
* Use of systemic retinoids (e.g isotretinoin, acitretin, bexarotene) within six months prior to study entry
* Within four weeks prior to study entry, use of acid containing products (e.g salicylic acids or fruit acids such as alpha and beta hydroxy acids and glycolic acids). located within 10 cm of the actinic keratosis lesion selected for treatment
* Anticipated need to use acid containing products on the treatment area during the study ( e.g salicylic acids or fruit acids, such as alpha and beta hydroxy acids and glycolic acids)
* Concurrent disease that supresses the immune system(e.g HIV)
* Uncontrolled systemic disease (e.g uncontrolled hypertension)
* Anticipated need for surgery or hospitalization during the study
* Current evidence of chronic alcohol or drug abuse
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Patient has a condition or is in a situation which in the Investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patients participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)

SECONDARY OUTCOMES:
Safety and clinical efficacy
Systemic absorption

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Anderson, MD, F.A.C.P, Principal Investigator
Locations (1):
- Dermatology Associates of Tyler, Tyler, Texas, United States